CLINICAL TRIAL: NCT05555173
Title: IVs With Buzzy in Chronic Pain Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left the institution
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 00838
Record Dates: First submitted 2022-09-16; First posted 2022-09-26 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Chronic Pain; Acute Pain
MeSH Terms: conditions — Chronic Pain; Acute Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Buzzy (Experimental): Buzzy will be applied 5 to 10 cm proximal (toward the subject's head) to the dorsum of the hand site immediately prior and throughout the intravenous catheter insertion attempt.
  Interventions: Device: Buzzy
- No Buzzy (No Intervention): Subjects will have a 20g intravenous catheter inserted either in the left or right dorsum side of the hand without the Buzzy device.

INTERVENTIONS:
Device: Buzzy — Buzzy is a small vibrating bee with ice-pack wings.
  Arms: Buzzy

SUMMARY:
The investigators are conducting a study to compare the effectiveness of the Buzzy® device with that of no pain relief method for IV placement in adults with chronic pain receiving lidocaine infusions.

DETAILED DESCRIPTION:
IV placement is necessary for lidocaine infusions. Unfortunately, some patients say that placing an IV is painful. The investigators are conducting this study to evaluate two techniques that could make the placement of the IV more comfortable. Currently, some medical providers administer the IV without any pain-relieving techniques. Some medical providers place a device called Buzzy® on a patient's arm prior to the IV placement. The Buzzy® device is the combination of an ice pack and a vibrator in the shape of a bumble bee. Literature shows that the Buzzy® device makes IV placement more comfortable for children, but there is minimal data in regard to whether it is helpful for adult patients. The investigators are conducting this study to compare the effectiveness of the Buzzy® device with that of no pain relief method for IV placement in adults with chronic pain receiving lidocaine infusions. The use of the Buzzy® device in adults is the investigational part of the study. This device has been FDA approved for use.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving lidocaine infusions at the pain clinic.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Pain on the Numeric Rating Scale | through study completion, an average of 2 months
  Patients are asked to report their subjective pain on the Numeric Rating Scale from 0 to 10, where 0 = No Pain and 10 = Worst Pain.

SECONDARY OUTCOMES:
Satisfaction on the Visual Analog Scale | through study completion, an average of 2 months
  Patients are asked to report their subjective satisfaction with the IV placement on the Visual Analog Scale, where labeled face images represent satisfaction from very poor satisfaction to excellent satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Gerges, MD, Principal Investigator — Pain Medicine Physician
Locations (1):
- St. Elizabeth's Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No